CLINICAL TRIAL: NCT04073719
Title: Apple Cider Vinegar for the Prevention of Urinary Lithiasis (APUL)
Acronym: APUL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christine Herforth, Urology Resident, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NMCSD.2019.0026
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Kidney Stones, Urolithiasis, Hypocitraturia
Keywords: Kidney Stones, Urolithiasis, Hypocitraturia, Apple Cider Vinegar
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Intervention Model Description: Prospective randomized sample of 36 patients, in a nested cross over design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Apple Cider Vinegar + Coconut Water (Experimental): Patients will drink apple cider vinegar for 7 days. After a washout period of 2 weeks, patients will then drink coconut water for 7 days.
  Interventions: Dietary Supplement: Apple Cider Vinegar
- Apple Cider Vinegar + Citric Soda (Experimental): Patients will drink apple cider vinegar for 7 days. After a washout period of 2 weeks, patients will then drink citric soda for 7 days.
  Interventions: Dietary Supplement: Apple Cider Vinegar
- Apple Cider Vinegar + Lemonade (Experimental): Patients will drink apple cider vinegar for 7 days. After a washout period of 2 weeks, patients will then drink lemonade for 7 days.
  Interventions: Dietary Supplement: Apple Cider Vinegar
- Coconut Water + Apple Cider Vinegar (Experimental): Patients will drink coconut water for 7 days. After a washout period of 2 weeks, patients will then drink apple cider vinegar for 7 days.
  Interventions: Dietary Supplement: Apple Cider Vinegar
- Coconut Water + Citric Soda (Experimental): Patients will drink coconut water for 7 days. After a washout period of 2 weeks, patients will then drink citric soda for 7 days.
  Interventions: Dietary Supplement: Other Beverage
- Coconut Water + Lemonade (Experimental): Patients will drink coconut water for 7 days. After a washout period of 2 weeks, patients will then drink lemonade for 7 days.
  Interventions: Dietary Supplement: Other Beverage
- Citric Soda + Apple Cider Vinegar (Experimental): Patients will drink citric soda for 7 days. After a washout period of 2 weeks, patients will then drink apple cider vinegar for 7 days.
  Interventions: Dietary Supplement: Apple Cider Vinegar; Dietary Supplement: Other Beverage
- Citric Soda + Coconut Water (Experimental): Patients will drink citric soda for 7 days. After a washout period of 2 weeks, patients will then drink coconut water for 7 days.
  Interventions: Dietary Supplement: Other Beverage
- Citric Soda + Lemonade (Experimental): Patients will drink citric soda for 7 days. After a washout period of 2 weeks, patients will then drink lemonade for 7 days.
  Interventions: Dietary Supplement: Other Beverage
- Lemonade + Apple Cider Vinegar (Experimental): Patients will drink lemonade for 7 days. After a washout period of 2 weeks, patients will then drink apple cider vinegar for 7 days.
  Interventions: Dietary Supplement: Apple Cider Vinegar
- Lemonade + Coconut Water (Experimental): Patients will drink lemonade for 7 days. After a washout period of 2 weeks, patients will then drink coconut water for 7 days.
  Interventions: Dietary Supplement: Other Beverage
- Lemonade + Citric Soda (Experimental): Patients will drink lemonade for 7 days. After a washout period of 2 weeks, patients will then drink citric soda for 7 days.
  Interventions: Dietary Supplement: Other Beverage

INTERVENTIONS:
Dietary Supplement: Apple Cider Vinegar — Will drinking apple cider vinegar increase urinary citrate levels to a greater degree than other beverages and which beverages produce the most significant effects compared against one another.
  Arms: Apple Cider Vinegar + Citric Soda; Apple Cider Vinegar + Coconut Water; Apple Cider Vinegar + Lemonade; Citric Soda + Apple Cider Vinegar; Coconut Water + Apple Cider Vinegar; Lemonade + Apple Cider Vinegar
Dietary Supplement: Other Beverage — To what degree do other high citrate beverages impact urinary citrate output.
  Arms: Citric Soda + Apple Cider Vinegar; Citric Soda + Coconut Water; Citric Soda + Lemonade; Coconut Water + Citric Soda; Coconut Water + Lemonade; Lemonade + Citric Soda; Lemonade + Coconut Water

SUMMARY:
The purpose of this study is to assess whether certain beverages can increase urinary citrate levels in healthy individuals with no history of kidney disease.

DETAILED DESCRIPTION:
Higher urinary citrate levels have been shown to decrease one's risk of developing kidney stones. The study will compare apple cider vinegar, coconut water, diet citric soda and lemonade and determine which is superior at raising citrate levels. Research participants will consume two of the four drinks, each for 7 day periods, according to a prescribed regimen. Throughout the course of the study, participants will periodically provide blood draws for metabolic panels, as well as 24-hour urine samples to measure citrate levels. There will be 12 study arms, accounting for the permutations of two drinks for each patients out of four possibilities. 3 participants per arm is the goal, for a total of 36, but the recruitment aim is 50 participants, to account for dropout and noncompliance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 18-65 years old

Exclusion Criteria:

* History of peptic ulcer disease or gastroparesis
* Pregnant females
* History of chronic kidney disease
* History of urolithiasis
* Currently taking medications that interfere with urinary electrolyte excretion (thiazide and loop diuretics)javascript:document.
* History of Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Apple Cider Vinegar Urinary Citrate Increase | 1 week
  Determine the change in urinary citrate levels due to the addition of apple cider vinegar to the diet

SECONDARY OUTCOMES:
Apple Cider Vinegar and urinary pH | 1 week
  Determine the effect of apple cider vinegar on urinary pH
Apple Cider Vinegar Against Other Beverages | 4 weeks
  Compare the effect of apple cider vinegar on urinary citrate with that of known citrate-rich beverages (lemonade, citrus based soda, coconut water)
Palatability Evaluation | 4 weeks
  Compare the palatability of apple cider vinegar and other known citrate-rich beverages (lemonade, citrus based soda, coconut water). Patients will keep daily log whwere they can free write any side effects (from palatability perspective and otherwise). At the end of the study a 2 question survery (Likert scale format) will be filled in which participants will answer the liklihood of their willingness to consume the beverage daily for the prevention of kidney stones.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Pearle MS, Calhoun EA, Curhan GC; Urologic Diseases of America Project. Urologic diseases in America project: urolithiasis. J Urol. 2005 Mar;173(3):848-57. doi: 10.1097/01.ju.0000152082.14384.d7. PMID 15711292
- [Background] Johnson CM, Wilson DM, O'Fallon WM, Malek RS, Kurland LT. Renal stone epidemiology: a 25-year study in Rochester, Minnesota. Kidney Int. 1979 Nov;16(5):624-31. doi: 10.1038/ki.1979.173. PMID 548606
- [Background] Bansal AD, Hui J, Goldfarb DS. Asymptomatic nephrolithiasis detected by ultrasound. Clin J Am Soc Nephrol. 2009 Mar;4(3):680-4. doi: 10.2215/CJN.05181008. Epub 2009 Mar 4. PMID 19261817
- [Background] Bhatti UH, Duffy AJ, Roberts KE, Shariff AH. Nephrolithiasis after bariatric surgery: A review of pathophysiologic mechanisms and procedural risk. Int J Surg. 2016 Dec;36(Pt D):618-623. doi: 10.1016/j.ijsu.2016.11.025. Epub 2016 Nov 12. PMID 27847289
- [Background] Maalouf NM, Tondapu P, Guth ES, Livingston EH, Sakhaee K. Hypocitraturia and hyperoxaluria after Roux-en-Y gastric bypass surgery. J Urol. 2010 Mar;183(3):1026-30. doi: 10.1016/j.juro.2009.11.022. Epub 2010 Jan 21. PMID 20096421
- [Background] Sakhaee K. Nephrolithiasis as a systemic disorder. Curr Opin Nephrol Hypertens. 2008 May;17(3):304-9. doi: 10.1097/MNH.0b013e3282f8b34d. PMID 18408483
- [Background] Sakhaee K, Maalouf NM, Kumar R, Pasch A, Moe OW. Nephrolithiasis-associated bone disease: pathogenesis and treatment options. Kidney Int. 2011 Feb;79(4):393-403. doi: 10.1038/ki.2010.473. Epub 2010 Dec 1. PMID 21124301
- [Background] Sakhaee K. Recent advances in the pathophysiology of nephrolithiasis. Kidney Int. 2009 Mar;75(6):585-95. doi: 10.1038/ki.2008.626. Epub 2008 Dec 10. PMID 19078968
- [Background] Worcester EM, Coe FL. Clinical practice. Calcium kidney stones. N Engl J Med. 2010 Sep 2;363(10):954-63. doi: 10.1056/NEJMcp1001011. No abstract available. PMID 20818905
- [Background] Curhan GC, Taylor EN. 24-h uric acid excretion and the risk of kidney stones. Kidney Int. 2008 Feb;73(4):489-96. doi: 10.1038/sj.ki.5002708. Epub 2007 Dec 5. PMID 18059457
- [Background] Nicar MJ, Skurla C, Sakhaee K, Pak CY. Low urinary citrate excretion in nephrolithiasis. Urology. 1983 Jan;21(1):8-14. doi: 10.1016/0090-4295(83)90113-9. PMID 6823713
- [Background] Rudman D, Kutner MH, Redd SC 2nd, Waters WC 4th, Gerron GG, Bleier J. Hypocitraturia in calcium nephrolithiasis. J Clin Endocrinol Metab. 1982 Dec;55(6):1052-7. doi: 10.1210/jcem-55-6-1052. PMID 7130336
- [Background] Pak CY, Poindexter JR, Adams-Huet B, Pearle MS. Predictive value of kidney stone composition in the detection of metabolic abnormalities. Am J Med. 2003 Jul;115(1):26-32. doi: 10.1016/s0002-9343(03)00201-8. PMID 12867231
- [Background] Pak CY. Citrate and renal calculi: an update. Miner Electrolyte Metab. 1994;20(6):371-7. PMID 7783699
- [Background] Zuckerman JM, Assimos DG. Hypocitraturia: pathophysiology and medical management. Rev Urol. 2009 Summer;11(3):134-44. PMID 19918339
- [Background] Ryall RL. Urinary inhibitors of calcium oxalate crystallization and their potential role in stone formation. World J Urol. 1997;15(3):155-64. doi: 10.1007/BF02201852. No abstract available. PMID 9228722
- [Background] Sheng X, Jung T, Wesson JA, Ward MD. Adhesion at calcium oxalate crystal surfaces and the effect of urinary constituents. Proc Natl Acad Sci U S A. 2005 Jan 11;102(2):267-72. doi: 10.1073/pnas.0406835101. Epub 2004 Dec 29. PMID 15625112
- [Background] Kok DJ, Papapoulos SE, Bijvoet OL. Excessive crystal agglomeration with low citrate excretion in recurrent stone-formers. Lancet. 1986 May 10;1(8489):1056-8. doi: 10.1016/s0140-6736(86)91329-2. PMID 2871335
- [Background] Preminger GM, Sakhaee K, Skurla C, Pak CY. Prevention of recurrent calcium stone formation with potassium citrate therapy in patients with distal renal tubular acidosis. J Urol. 1985 Jul;134(1):20-3. doi: 10.1016/s0022-5347(17)46963-1. PMID 4009822
- [Background] Pak CY, Fuller C, Sakhaee K, Preminger GM, Britton F. Long-term treatment of calcium nephrolithiasis with potassium citrate. J Urol. 1985 Jul;134(1):11-9. doi: 10.1016/s0022-5347(17)46962-x. PMID 3892044
- [Background] Pak CY, Sakhaee K, Fuller C. Successful management of uric acid nephrolithiasis with potassium citrate. Kidney Int. 1986 Sep;30(3):422-8. doi: 10.1038/ki.1986.201. PMID 3784284
- [Background] Barcelo P, Wuhl O, Servitge E, Rousaud A, Pak CY. Randomized double-blind study of potassium citrate in idiopathic hypocitraturic calcium nephrolithiasis. J Urol. 1993 Dec;150(6):1761-4. doi: 10.1016/s0022-5347(17)35888-3. PMID 8230497
- [Background] Ettinger B, Pak CY, Citron JT, Thomas C, Adams-Huet B, Vangessel A. Potassium-magnesium citrate is an effective prophylaxis against recurrent calcium oxalate nephrolithiasis. J Urol. 1997 Dec;158(6):2069-73. doi: 10.1016/s0022-5347(01)68155-2. PMID 9366314
- [Background] Soygur T, Akbay A, Kupeli S. Effect of potassium citrate therapy on stone recurrence and residual fragments after shockwave lithotripsy in lower caliceal calcium oxalate urolithiasis: a randomized controlled trial. J Endourol. 2002 Apr;16(3):149-52. doi: 10.1089/089277902753716098. PMID 12028622
- [Background] Kang DE, Maloney MM, Haleblian GE, Springhart WP, Honeycutt EF, Eisenstein EL, Marguet CG, Preminger GM. Effect of medical management on recurrent stone formation following percutaneous nephrolithotomy. J Urol. 2007 May;177(5):1785-8; discussion 1788-9. doi: 10.1016/j.juro.2007.01.061. PMID 17437820
- [Background] Mattle D, Hess B. Preventive treatment of nephrolithiasis with alkali citrate--a critical review. Urol Res. 2005 May;33(2):73-9. doi: 10.1007/s00240-005-0464-8. Epub 2005 May 4. PMID 15875173
- [Background] Koff SG, Paquette EL, Cullen J, Gancarczyk KK, Tucciarone PR, Schenkman NS. Comparison between lemonade and potassium citrate and impact on urine pH and 24-hour urine parameters in patients with kidney stone formation. Urology. 2007 Jun;69(6):1013-6. doi: 10.1016/j.urology.2007.02.008. PMID 17572176
- [Background] Seltzer MA, Low RK, McDonald M, Shami GS, Stoller ML. Dietary manipulation with lemonade to treat hypocitraturic calcium nephrolithiasis. J Urol. 1996 Sep;156(3):907-9. PMID 8709360
- [Background] Kang DE, Sur RL, Haleblian GE, Fitzsimons NJ, Borawski KM, Preminger GM. Long-term lemonade based dietary manipulation in patients with hypocitraturic nephrolithiasis. J Urol. 2007 Apr;177(4):1358-62; discussion 1362; quiz 1591. doi: 10.1016/j.juro.2006.11.058. PMID 17382731
- [Background] Penniston KL, Steele TH, Nakada SY. Lemonade therapy increases urinary citrate and urine volumes in patients with recurrent calcium oxalate stone formation. Urology. 2007 Nov;70(5):856-60. doi: 10.1016/j.urology.2007.06.1115. Epub 2007 Oct 24. PMID 17919696
- [Background] Odvina CV. Comparative value of orange juice versus lemonade in reducing stone-forming risk. Clin J Am Soc Nephrol. 2006 Nov;1(6):1269-74. doi: 10.2215/CJN.00800306. Epub 2006 Aug 30. PMID 17699358
- [Background] Penniston KL, Nakada SY, Holmes RP, Assimos DG. Quantitative assessment of citric acid in lemon juice, lime juice, and commercially-available fruit juice products. J Endourol. 2008 Mar;22(3):567-70. doi: 10.1089/end.2007.0304. PMID 18290732
- [Background] Haleblian GE, Leitao VA, Pierre SA, Robinson MR, Albala DM, Ribeiro AA, Preminger GM. Assessment of citrate concentrations in citrus fruit-based juices and beverages: implications for management of hypocitraturic nephrolithiasis. J Endourol. 2008 Jun;22(6):1359-66. doi: 10.1089/end.2008.0069. PMID 18578663
- [Background] Patel RM, Jiang P, Asplin J, Granja I, Capretz T, Osann K, Okhunov Z, Landman J, Clayman RV. Coconut Water: An Unexpected Source of Urinary Citrate. Biomed Res Int. 2018 Nov 1;2018:3061742. doi: 10.1155/2018/3061742. eCollection 2018. PMID 30515390
- [Background] Yamashita H. Biological Function of Acetic Acid-Improvement in Obesity and Glucose Tolerance by Acetic Acid in Type 2 Diabetic Rats. Crit Rev Food Sci Nutr. 2016 Jul 29;56 Suppl 1:S171-5. doi: 10.1080/10408398.2015.1045966. PMID 26176799
- [Background] Yamashita H, Fujisawa K, Ito E, Idei S, Kawaguchi N, Kimoto M, Hiemori M, Tsuji H. Improvement of obesity and glucose tolerance by acetate in Type 2 diabetic Otsuka Long-Evans Tokushima Fatty (OLETF) rats. Biosci Biotechnol Biochem. 2007 May;71(5):1236-43. doi: 10.1271/bbb.60668. Epub 2007 May 7. PMID 17485860
- [Background] Kondo T, Kishi M, Fushimi T, Ugajin S, Kaga T. Vinegar intake reduces body weight, body fat mass, and serum triglyceride levels in obese Japanese subjects. Biosci Biotechnol Biochem. 2009 Aug;73(8):1837-43. doi: 10.1271/bbb.90231. Epub 2009 Aug 7. PMID 19661687
- [Background] Brighenti F, Castellani G, Benini L, Casiraghi MC, Leopardi E, Crovetti R, Testolin G. Effect of neutralized and native vinegar on blood glucose and acetate responses to a mixed meal in healthy subjects. Eur J Clin Nutr. 1995 Apr;49(4):242-7. PMID 7796781
- [Background] White AM, Johnston CS. Vinegar ingestion at bedtime moderates waking glucose concentrations in adults with well-controlled type 2 diabetes. Diabetes Care. 2007 Nov;30(11):2814-5. doi: 10.2337/dc07-1062. Epub 2007 Aug 21. No abstract available. PMID 17712024
- [Background] Johnston CS, Kim CM, Buller AJ. Vinegar improves insulin sensitivity to a high-carbohydrate meal in subjects with insulin resistance or type 2 diabetes. Diabetes Care. 2004 Jan;27(1):281-2. doi: 10.2337/diacare.27.1.281. No abstract available. PMID 14694010
- [Background] Shishehbor F, Mansoori A, Sarkaki AR, Jalali MT, Latifi SM. Apple cider vinegar attenuates lipid profile in normal and diabetic rats. Pak J Biol Sci. 2008 Dec 1;11(23):2634-8. doi: 10.3923/pjbs.2008.2634.2638. PMID 19630216
- [Derived] Baker B, Herforth C, Low J, Craig R, Christman M. Apple cider vinegar for prevention of urinary lithiasis (APUL): a randomized crossover trial. Int Urol Nephrol. 2025 Dec 6. doi: 10.1007/s11255-025-04944-x. Online ahead of print. PMID 41351751